CLINICAL TRIAL: NCT02796521
Title: Evaluation of the Effectiveness of Nutritional Practical Counseling for Elderly Patients at Risk of Malnutrition (and Their Caregivers) on Nutritional Status at Home
Brief Title: Evaluation of Effectiveness of Nutritional Practical Counseling for Elderly Patients at Risk of Malnutrition on Nutritional Status at Home
Acronym: NutriPratiC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no more budget for personal to enrol participants
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 38RC14.177
Record Dates: First submitted 2016-06-01; First posted 2016-06-10 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2016-05

CONDITIONS: Malnutrition
Keywords: malnutrition; aging; diet therapy
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Other): The control group will receive usual dietary counseling for enrichment.
  Interventions: Other: dietary counseling
- workshop group (Other): The workshop group will have informations about interest of foods. They will enrich a meal with foods which can easily be added without cooking.
  Interventions: Other: dietary counseling; Other: nutritional workshop with enrichment during a meal

INTERVENTIONS:
Other: dietary counseling — Patients received individualized nutritional counseling encouraging them for enrichment
Other: nutritional workshop with enrichment during a meal — Patients received in group nutritional informations for enrichment and are encouraged to try enrichment together during a meal.
  Arms: workshop group

SUMMARY:
At hospital, short term actions are used (adaptation of meals, oral supplementation…) to fight malnutrition. Oral supplementation can have a positive impact on weight gain. But actions should continue at home, particularly to maintain autonomy for elderly. The hypothesis is that practical workshop about enrichment and interest of foods can help malnourished patients to change their eating habits. The main goal of this study is to evaluate the effects of this workshop on improving nutritional status, measured by Mini Nutritional Assessment

DETAILED DESCRIPTION:
This is a mono center cohort study of a 4-months follow-up on elderly patients after hospitalization.

Nutritional parameters and evaluation of the quality of life will be collected during hospitalization and output during a visit at 4 months at home. These parameters will be studied in two groups : nutritional workshop vs usual dietary counseling

ELIGIBILITY:
Inclusion Criteria:

* malnourished patients or at risk of malnutrition
* coming back home after hospitalization
* affiliated to a social security system
* having given free, informed written consent

Exclusion Criteria:

* Mini Mental Score <18
* Incapacitated adults and psychiatric inpatients
* Diet indication requiring strict salt restriction
* Severe swallowing difficulties
* Patients with artificial nutrition (enteral or parenteral)
* Impossibility to measure weight at home
* Severe digestive or intestinal malabsorption
* Iterative nausea and vomiting
* Patients with rapidly progressive diseases (life expectancy less than 6 months)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Improvement of nutritional status | 4 months
  global Mini Nutritional Assessment

SECONDARY OUTCOMES:
Effect of the workshop on nutritional items of Mini Nutritional Assessment | 4 months
  specific nutritional items of Mini Nutritional Assessment
Maintaining or improving weight | 4 months
  Weight is determined with a Seca floor scale
Improving ingesta qualitatively and quantitatively | 4 months
  Ingesta are determined with a 24h-recall questionnaire
Representations and motivations on eating habits | 4 months
  Representations and motivations on eating habits are determined with a questionnaire with Likert responses
Rate returns to the hospital and not programmed planned | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnaud-Battandier F, Malvy D, Jeandel C, Schmitt C, Aussage P, Beaufrere B, Cynober L. Use of oral supplements in malnourished elderly patients living in the community: a pharmaco-economic study. Clin Nutr. 2004 Oct;23(5):1096-103. doi: 10.1016/j.clnu.2004.02.007. PMID 15380901
- [Background] Boumendjel N, Herrmann F, Girod V, Sieber C, Rapin CH. Refrigerator content and hospital admission in old people. Lancet. 2000 Aug 12;356(9229):563. doi: 10.1016/S0140-6736(00)02583-6. PMID 10950235
- [Background] Correia MI, Waitzberg DL. The impact of malnutrition on morbidity, mortality, length of hospital stay and costs evaluated through a multivariate model analysis. Clin Nutr. 2003 Jun;22(3):235-9. doi: 10.1016/s0261-5614(02)00215-7. PMID 12765661
- [Background] McMurdo ME, Price RJ, Shields M, Potter J, Stott DJ. Should oral nutritional supplementation be given to undernourished older people upon hospital discharge? A controlled trial. J Am Geriatr Soc. 2009 Dec;57(12):2239-45. doi: 10.1111/j.1532-5415.2009.02568.x. Epub 2009 Nov 17. PMID 19925613
- [Background] Persson M, Hytter-Landahl A, Brismar K, Cederholm T. Nutritional supplementation and dietary advice in geriatric patients at risk of malnutrition. Clin Nutr. 2007 Apr;26(2):216-24. doi: 10.1016/j.clnu.2006.12.002. Epub 2007 Feb 1. PMID 17275141
- [Background] Ravasco P, Monteiro-Grillo I, Vidal PM, Camilo ME. Dietary counseling improves patient outcomes: a prospective, randomized, controlled trial in colorectal cancer patients undergoing radiotherapy. J Clin Oncol. 2005 Mar 1;23(7):1431-8. doi: 10.1200/JCO.2005.02.054. Epub 2005 Jan 31. PMID 15684319